CLINICAL TRIAL: NCT05063669
Title: Effects of Cognitive Occupational Therapy Interventions on Executive Functions in Children With Attention Deficit and Hyperactivity Disorder
Brief Title: Cognitive Intervention in Attention Deficit and Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Remziye Akarsu, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniOccupationalTherapy
Record Dates: First submitted 2021-09-15; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: ADHD; Cognitive Deficit
Keywords: Attention Deficit and Hyperactivity Disorder; Executive functions; Occupational therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Occupational Therapy (Experimental): Occupational therapy applications were carried out 40 minutes, twice a week (one individual session and one group intervention session) and total of 8 weeks. In the sessions, activities aimed at reasoning and empathy skills, problem solving, evaluating emotional cues, evaluating events from different perspectives, providing personal control, delaying reactions, motor planning, visual perception and prolonging attention span were applied. The interventions were varied according to the personal characteristics of the individuals. In group interventions with three or four participants, group games in the form of cooperation or competition were planned to develop motor planning and cognitive strategy and it was aimed to improve children's rapid decision making and adaptation skills.
  Interventions: Behavioral: Cognitive Occupational Therapy
- Control (No Intervention): No intervention was performed in this group.

INTERVENTIONS:
Behavioral: Cognitive Occupational Therapy — In the sessions, activities aimed at reasoning and empathy skills, problem solving, evaluating emotional cues, evaluating events from different perspectives, providing personal control, delaying reactions, motor planning, visual perception and prolonging attention span were applied. The interventions were varied according to the personal characteristics of the individuals. In group interventions with three or four participants, group games in the form of cooperation or competition were planned to develop motor planning and cognitive strategy and it was aimed to improve children's rapid decision making and adaptation skills.
  Arms: Cognitive Occupational Therapy

SUMMARY:
Attention Deficit Hyperactivity Disorder is a disorder in which children show insufficient attention span, hyperactivity and impulsivity according to their developmental level. It is stated that in the absence of rehabilitation, the child's social and academic functionality gradually deteriorates, there are problems in cognitive function processes and executive dysfunctions that affect daily life. The aim of this study was to investigate the effects of cognitive occupational therapy interventions on executive functions in children with Attention Deficit and Hyperactivity Disorder. 21 children aged 9-12 years were included in the research (10 study group-11 control group). One individual and one group session was applied to the study group at Biruni University Occupational Therapy Unit as 2 times per week for 8 weeks. Both groups were evaluated at the beginning and after 8 weeks with Children's Color Trails Test, Verbal Fluency Test and Stroop Test T-Bag Form. Wilcoxon Paired Sample Test and Mann Whitney U Test were used for analysis of intervention results and comparison between groups.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a neuropsychiatric disorder marked by an ongoing pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or growing. In individuals with ADHD, clinical findings may vary depending on development. It is frequently observed that ADHD, which has a progressive character, continues into adulthood after childhood and adolescence.

The study was conducted in Biruni University Occupational Therapy Unit. Since the individuals participating in the study were under the age of 18, an informed consent form was signed by their parents. The research was carried out between June and December 2020. The study included children aged 9-12 years who were diagnosed with ADHD according to DSM-V criteria by a psychiatrist, did not use any medication for ADHD, or were given a fixed dose 3 months ago and did not plan to change their treatment. Children who could not participate in the study because of any medical or mental health problems and who were diagnosed with any secondary diagnosis were excluded. First of all, the sociodemographic form was applied to the participants. The form consisted of questions to determine age, gender, disease history, presence of drugs used continuously, education level of parents, and whether the participant or family member had neurological or psychiatric disorders. Stroop Test T Bag Form (ST-TBAG), The Children's Color Trails Test (CCTT) and Verbal Fluency Test (VFT) were applied to all participants before and after intervention. Occupational therapy applications were carried out 40 minutes, twice a week (one individual session and one group intervention session) and total of 8 weeks. In the sessions, activities aimed at reasoning and empathy skills, problem solving, evaluating emotional cues, evaluating events from different perspectives, providing personal control, delaying reactions, motor planning, visual perception and prolonging attention span were applied. The interventions were varied according to the personal characteristics of the individuals. In group interventions with three or four participants, group games in the form of cooperation or competition were planned to develop motor planning and cognitive strategy and it was aimed to improve children's rapid decision making and adaptation skills.

Research data were evaluated in SPSS 22.0 package program. Mean±standard deviation (X±SD) was determined for the variables determined by measurement. The Wilcoxon Paired Two-Sample Test was used to compare the first and last evaluation data of the intervention and control groups and the Mann Whitney-U test was used to compare the demographic and initial evaluation data of both groups. A significance value of p<0.05 was accepted in all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9-12 years
* Clinical diagnosis of ADHD according to DSM-V criteria by a psychiatrist
* Not taking any medication for ADHD or taking a fixed dose 3 months ago

Exclusion Criteria:

* Any medical or mental health problems
* Any secondary diagnosis

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Stroop Test T Bag Form | 2 weeks
  Stroop Test T Bag Form evaluates selective or focused attention and is administered with four 14x21.5 cm white cards. On the first card, random color names (blue, green, red, yellow) are printed in black letters, in a total of 10 rows with five words per line. The second card has the same number of dots printed with these colors, the third card has the same number of color names with the colors written (each written color name is printed in a different color), the fourth card has random words written in different colors.14 Participants were first asked to read the black printed card as fast as possible. The errors and corrections made during this period and the total time spent were recorded. Color names written in color in the second stage, the colors of the shapes in the third stage, word colors without color names in the fourth stage and in the fifth stage, the test was completed by recording the accuracy and duration of saying the word colors, which are the color names.
The Children's Color Trails Test | 2 weeks
  The Children's Color Trails Test was used as a measure in which the first part measures psychomotor speed and the second part evaluates executive function and visuospatial working memory, reflecting the ability to change strategy.
Verbal Fluency Test | 2 weeks
  Verbal Fluency Test VFT is a short screening test that evaluates cognitive function. The two most commonly used variations of the test focus on semantic and phonemic criteria.13 In the first, words in the same semantic field are requested (for example, animals), in the second, it is requested to evoke as many words with the same phoneme as possible (for example, words starting with /a/). One minute was determined for each letter (the letter B is given as an example) and the participant was asked to say every word that can be remembered, provided that there were no proper names starting with the letters K, A and S. Then they were asked to count the fruits, animals and products that could be bought in the supermarket, again for one minute per category and the results were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Remziye Akarsu, MS, Principal Investigator — Biruni University; Başar Öztürk, PhD, Study Director — Biruni University; Amine Karademir, Bachelor, Study Chair — Biruni University; Melek Görgülü, Bachelor, Study Chair — Biruni University; Betül Güler, Bachelor, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No